CLINICAL TRIAL: NCT03209804
Title: Surgical Management of Cerebral Arteriovenous Malformations Within Hybrid Operation Room
Acronym: SMAVMHR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Shuo Wang, liuxingju, Beijing Tiantan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BJTTH-002
Record Dates: First submitted 2017-06-26; First posted 2017-07-06 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Intracranial Arteriovenous Malformations
Keywords: Intracranial Arteriovenous Malformations
MeSH Terms: conditions — Intracranial Arteriovenous Malformations

STUDY DESIGN:
Intervention Model Description: Traditional therapy group：traditional management of AVMs, such as unsimultaneous endovascular interventional embolisation, radiotherapy followed by microsurgical resection, will be conducted to patients involved in this group.
  Hybrid operation group: A one-stage hybrid operation combining endovascular intervention and microsurgical techniques will be conducted simultaneously to patients in this group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional neurosurgical techniques (Other): Unsimultaneous endovascular interventional embolisation/radiotherapy followed by microsurgical resection, as traditional clinical routines.
  Interventions: Procedure: hybrid operating techniques
- Hybrid operating techniques (Experimental): A one-stage hybrid operation combining endovascular intervention and microsurgical techniques will be conducted simultaneously
  Interventions: Procedure: hybrid operating techniques

INTERVENTIONS:
Procedure: hybrid operating techniques — A one-stage cooperation of existing endovascular interventional techniques and microsurgical techniques, including microsurgical resection, endovascular embolization, balloon occlusion.
  Other Names: endovascular interventional embolisation; endovascular interventional balloon occlusion; microsurgical resection

SUMMARY:
To evaluate the clinical benefits and risks of hybrid operating techniques in management of cerebral arteriovenous malformations.

DETAILED DESCRIPTION:
Purpose: Have an evaluation of clinical benefits and risks of hybrid operating techniques in management of cerebral arteriovenous malformations(AVMs). Meanwhile, as a new cooperative interventional modality, optimized workflows, technical key knots and operation routines will be explored in the study.

Objects: Patients with cerebral arteriovenous malformations, coincident with inclusion and exclusion criterion and admitted in participating organizations.

Methods: Patients will be distributed into 2 groups, including traditional therapy group(control group) and hybrid operating group(trial group), and conduct with traditional neurosurgical management or one-stage hybrid operating management correspondingly. Residual rate of AVM is considered to be the primary observing indicator, and morbidity rate of post-operative complications, post-operative mortality rate, and morbidity rate of neural functional deterioration are secondary indicators.The information of operations will be recorded in detail as evidence of optimization of workflow and technical key knots.

ELIGIBILITY:
Inclusion Criteria:

* newly ruptured AVM with stable hematoma, selective operation is practical;
* with rupture history;
* recurrent epilepsy, failed in AED management;
* giant AVM with deterioration of neurological functions;
* 1-4 grade AVM (Spetzler-Martin grading system) with no symptom and not located in eloquent area.

Exclusion Criteria:

* >70 in age, with low rupture risk;
* newly ruptured AVM with unstable hematoma, engaged in emergency operation;
* ≥5 grade in Spetzler-Martin grading system;
* AVM located in hypothalamus, brainstem, cerebellopontine angle;
* cannot tolerant the operation;
* patient or relative refuses to participate the trail.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2016-06; Primary Completion 2019-12 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Instant residual rate of AVMs | up to 1 week after operation
  The instant post-operative residual rate of AVMs
3 months' residual rate of AVMs | the date of 3rd month after operation, ±1 week
  3 months' residual rate after AVM operation
6 months' residual rate of AVMs | the date of the 6th month after operation, ±1 week
  6 months' residual rate after AVM operation
1 year's residual rate of AVMs | the date of the 12th month after operation, ±1 week
  1 year's residual rate after AVM operation

SECONDARY OUTCOMES:
Morbidity rate of post-operative complications | 7 days after operation
  Include intracranial hemorrhage or infarction, infection of central neural system, infection of respiratory system, cranial nerve deficits, and other symptomatic complications
Post-operative mortality rate | 48 hours after operation
  operation related mortality
Morbidity rate of neural functional deterioration-48 hours after operation | the assessing time points is 48 hours after operation
  The score of modified Rankin Scale increases ≥2
Morbidity rate of neural functional deterioration-1 week after operation | 1 week after operation
  The score of modified Rankin Scale increases ≥2
Morbidity rate of neural functional deterioration-3 months after operation | the 3rd month after operation, ±1 week
  The score of modified Rankin Scale increases ≥2
Morbidity rate of neural functional deterioration-6 months after operation | the 6th month after operation, ±1 week
  The score of modified Rankin Scale increases ≥2
Morbidity rate of neural functional deterioration-12 months after operation | the 12th month after operation, ±1 week
  The score of modified Rankin Scale increases ≥2

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Beijing Tiantan Hospital Capital Medical University, Beijing, Beijing Municipality
  - General Hospital of PLA, Beijing, Beijing Municipality
  - Rocket Army General Hospital of PLA, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided